CLINICAL TRIAL: NCT00652106
Title: Safety and Efficacy Study of Brimonidine/Timolol Fixed Combination in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190342-019T
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination; Timolol; Ophthalmic Solutions; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): 0.2% brimonidine/0.5% timolol fixed combination ophthalmic solution
  Interventions: Drug: 0.2% brimonidine/0.5% timolol fixed combination ophthalmic solution
- 2 (Active Comparator): Concurrent brimonidine 0.2% and Timolol 0.5% ophthalmic solution
  Interventions: Drug: Concurrent brimonidine 0.2% and Timolol 0.5% ophthalmic solution
- 3 (Active Comparator): 0.2% brimonidine ophthalmic solution
  Interventions: Drug: Brimonidine 0.2% ophthalmic solution

INTERVENTIONS:
Drug: 0.2% brimonidine/0.5% timolol fixed combination ophthalmic solution — 0.2% brimonidine/0.5% timolol fixed combination ophthalmic solution 1 drop instilled in each eye twice daily (morning and evening)
  Other Names: COMBIGAN®
  Arms: 1
Drug: Concurrent brimonidine 0.2% and Timolol 0.5% ophthalmic solution — Brimonidine 0.2% 1 drop instilled in each eye three times daily (morning, afternoon, and evening) and concurrent timolol 0.5% ophthalmic solution 1 drop instilled in each eye twice daily (morning and evening)
  Arms: 2
Drug: Brimonidine 0.2% ophthalmic solution — Brimonidine 0.2% ophthalmic solution 1 drop instilled in each eye three times daily (morning, afternoon, and evening)
  Other Names: ALPHAGAN®
  Arms: 3

SUMMARY:
This study evaluates the safety and efficacy of brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution compared with concurrent brimonidine 0.2% and timolol ophthalmic solutions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension or glaucoma
* Patient requires IOP-lowering therapy in both eyes

Exclusion Criteria:

* Uncontrolled medical conditions
* Contraindication to β-adrenoceptor antagonist therapy or brimonidine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2003-06; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- El Paso, Texas, United States

REFERENCES:
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com